CLINICAL TRIAL: NCT00444665
Title: Examining The Efficacy, Safety And Improved Tolerability Of Travoprost BAK Free Ophthalmic Solution (Travatan-Z) Compared To Prior Prostaglandin Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-06-24
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2008-04

CONDITIONS: Glaucoma
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Travoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Travatan-Z

SUMMARY:
Examine the safety, tolerability and efficacy of travoprost benzalkonium chloride (BAK) free ophthalmic solution compared to either latanoprost or bimatoprost monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a clinical diagnosis of ocular hypertension, or primary open-angle, pigment dispersion or exfoliation glaucoma in at least one eye (study eye)

Exclusion Criteria:

* Age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2007-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Symptoms

SECONDARY OUTCOMES:
Intraocular pressure

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jasek, PhD, Study Director — Alcon Research
Locations (1):
- Fridley, Fridley, Minnesota, United States

REFERENCES:
- [Result] Henry JC, Peace JH, Stewart JA, Stewart WC. Efficacy, safety, and improved tolerability of travoprost BAK-free ophthalmic solution compared with prior prostaglandin therapy. Clin Ophthalmol. 2008 Sep;2(3):613-21. doi: 10.2147/opth.s3881. PMID 19668762